CLINICAL TRIAL: NCT00579436
Title: Effects of Fish Oils on Inflammation and Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Kern (Other)
Collaborators: GlaxoSmithKline (Industry); National Institutes of Health (NIH) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor-Investigator, Philip Kern, Professor of Medicine, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 74457; P20RR021954 (NIH)
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Results first posted 2018-05-16 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-04

CONDITIONS: Metabolic Syndrome; Insulin Resistance
Keywords: inflammation; obesity; diabetes
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance; Inflammation; Obesity; Diabetes Mellitus | interventions — Fatty Acids, Omega-3; Omacor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fish oil group (Active Comparator): 4g Lovaza (omega-3 fatty acid) daily.
  Interventions: Drug: omega-3 fatty acid
- Control group (Placebo Comparator): placebo (4 non-active capsules daily)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: omega-3 fatty acid — 4g of omega-3 fatty acid daily by mouth for 12 weeks.
  Other Names: Lovaza
  Arms: Fish oil group
Drug: placebo — 4 inert capsules daily by mouth for 12 weeks.
  Arms: Control group

SUMMARY:
The purpose of this study is to determine whether improvement in fat and muscle metabolism after the treatment with Omacor (fish oils) provides insight into the link between obesity, fat and muscle function leading to metabolic syndrome, which is a risk factor for heart disease and diabetes.

DETAILED DESCRIPTION:
The development of type 2 diabetes (T2DM) represents a complex series of events, involving abnormalities in adipose tissue lipid distribution and insulin action. Along with an increase in adipose tissue mass is an increase in inflammation brought about by macrophages that infiltrate adipose tissue. These macrophages express inflammatory cytokines such as tumor necrosis factor (TNF) and Interleukin -6 (IL-6) which are correlated with insulin resistance and metabolic syndrome, and suggest that metabolic syndrome and diabetes are conditions characterized by a state of chronic, low-grade inflammation. Thiazolidinediones (TZDs) improve insulin sensitivity via activation of peroxisome proliferator-activated receptor (PPAR) , and there is much evidence that PPAR agonists also have anti-inflammatory properties.

Fish oils are rich sources of Omega-3 fatty acids and there is a large literature on the potential benefits of fish oils on lowering serum triglycerides, cardiovascular protection, and immune modulation, and there is evidence that fish oils also activate PPAR . Hence, the focus of this study will be on subjects with insulin resistance and metabolic syndrome, but who do not yet have diabetes. We plan to treat insulin resistant subjects with fish oils and ask the following questions.

Hypothesis 1. The treatment of insulin resistant subjects with fish oils will reduce adipose tissue inflammation.

Aim 1. From blood samples drawn before and after treatment, we will measure levels of circulating inflammatory cytokines.

Aim 2. Adipose tissue biopsies will be performed before and after fish oil treatment. From the adipose biopsies, we will quantitate cytokine expression, macrophage number, and we will look for evidence of macrophage apoptosis.

Aim 3. We will determine whether fish oil treatment increases the adipose tissue secretion and serum level of the high molecular weight form of adiponectin.

Hypothesis 2. The reduction in inflammatory markers occurs through an activation of PPAR by the fish oils.

Aim 4. Adipose tissue and macrophages will be treated in vitro with fish oils in the presence and absence of a PPAR inhibitor. We will determine whether fish oils stimulate the secretion of the high molecular weight adiponectin isoform from adipose tissue and whether they induce apoptosis from macrophages, and whether this process is inhibited by the PPAR inhibitor.

Hypothesis 3. Fish oils improve peripheral insulin sensitivity through a reduction in intramyocellular lipid, and an improvement in muscle insulin signal transduction.

Aim 5. Before and after treatment with fish oils, insulin sensitivity will be measured, along with intramyocellular lipid and genes involved in insulin action and muscle lipid oxidation.

ELIGIBILITY:
Inclusion Criteria:

* BMI 27-45 kg/m2
* age 35-65 years
* abnormal carbohydrate metabolism

Exclusion Criteria:

* triglycerides over 700 mg/dl
* renal disease
* liver disease
* congestive heart failure
* history of heart disease or stroke
* chronic aspirin or NSAID use (anti-coagulant)
* history of a bleeding disorder
* use of statins, fibrates, ACE inhibitors, angiotensin II receptor blockers and glucocorticoids
* diet heavy in omega-3 fatty acids (salmon, sardines, flaxseeds)

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-01; Primary Completion 2013-03-27 (Actual); Study Completion 2015-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip A. Kern, M.D., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Medical Cener, Lexington, Kentucky, United States

REFERENCES:
- [Result] Spencer M, Finlin BS, Unal R, Zhu B, Morris AJ, Shipp LR, Lee J, Walton RG, Adu A, Erfani R, Campbell M, McGehee RE Jr, Peterson CA, Kern PA. Omega-3 fatty acids reduce adipose tissue macrophages in human subjects with insulin resistance. Diabetes. 2013 May;62(5):1709-17. doi: 10.2337/db12-1042. Epub 2013 Jan 17. PMID 23328126

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Non-diabetic subjects with either impaired glucose tolerance, impaired fasting glucose, or at least three features of metabolic syndrome were recruited at the University of Kentucky or the University of Arkansas. Exclusion criteria included history of coronary heart disease, inflammatory disease or chronic anti-inflammatory use
Period: Overall Study
Arm/Group | Fish Oil Group | Control Group
Started | 19 | 14
Completed | 19 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fish Oil Group | Control Group | Total
Number analyzed (Participants) | 19 | 14 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (9.8) | 53.3 (8.3) | 50.8 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United States | 19 | 14 | 33
Weight [Mean (Standard Deviation); unit: kilograms] | 99.8 (12.5) | 92.1 (16.9) | 96.8 (14.9)
Body fat [Mean (Standard Deviation); unit: percent] | 44.4 (7.4) | 46.2 (10.1) | 44.9 (8.64)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 33.4 (5.4) | 33.8 (4.3) | 33.4 (4.9)
Triglycerides [Mean (Standard Deviation); unit: mg/dl] | 150 (57.92) | 163.0 (82.8) | 155.7 (69)
Cholesterol [Mean (Standard Deviation); unit: mg/dl] | 207.1 (41.6) | 204.7 (44.5) | 206 (42.3)
High density lipoprotein [Mean (Standard Deviation); unit: mg/dl] | 53.5 (15.21) | 47.7 (12.2) | 49.50 (13.63)
Low density lipoprotein [Mean (Standard Deviation); unit: mg/dl] | 125.9 (36.8) | 122.4 (40.8) | 125.5 (37.5)
2 hour Glucose [Mean (Standard Deviation); unit: mg/dl] | 167.8 (43.3) | 157.8 (29.0) | 163.1 (37.6)
HbA1c [Mean (Standard Deviation); unit: percent] | 6.0 (.3) | 5.6 (0.4) | 5.8 (.4)

OUTCOME MEASURES:

1. Primary Outcome: Baseline Adipocyte Size
Description: Prior to starting the fish oil regiment, participants will undergo an incisional abdominal biopsy to remove approximately 4g of adipose tissue to determine adipocyte size
Time Frame: baseline
Measure: Mean (Standard Error); unit: square micrometers
Arm/Group | Fish Oil Group | Control Group
Number analyzed (Participants) | 19 | 14
square micrometers | 4958 (249) | 4489 (231)
Statistical Analysis 1: Comparison: Fish Oil Group vs Control Group; Test type: Superiority; p = .05, t-test, 2 sided

2. Primary Outcome: Adipocyte Size After Fish Oil Treatment
Description: After completing the fish oil regiment, participant will undergo an incisional abdominal biopsy to remove approximately 4g of adipose tissue to determine individual adipocyte size
Time Frame: week 12
Measure: Mean (Standard Error); unit: square micrometers
Arm/Group | Fish Oil Group | Control Group
Number analyzed (Participants) | 19 | 14
square micrometers | 4869 (209) | 4051 (191)
Statistical Analysis 1: Comparison: Fish Oil Group vs Control Group; Test type: Superiority; p = 0.05, t-test, 2 sided

3. Secondary Outcome: Baseline Insulin Resistance
Description: Insulin sensitivity (Si) was measured with a frequently sampled intravenous glucose tolerance test. Participants received a bolus of glucose at Time Zero, then a bolus of insulin 20 minutes later. Blood was collected through an IV catheter at multiple time points over the course of 4 hours. Glucose levels were plotted on a time course curve and analyzed using the MIDMOD algorithm.
Time Frame: baseline
Population: all participants were analyzed
Measure: Mean (Standard Error); unit: [mU/L]^-1 x [min]^-1]
Arm/Group | Fish Oil Group | Control Group
Number analyzed (Participants) | 19 | 14
[mU/L]^-1 x [min]^-1] | 1.8 (.2) | 1.8 (0.3)
Statistical Analysis 1: Comparison: Fish Oil Group vs Control Group; Test type: Superiority; p = 0.5, t-test, 2 sided

4. Secondary Outcome: Insulin Resistance After Fish Oil Regiment
Description: Insulin sensitivity (Si) was measured with a frequently sampled intravenous glucose tolerance test. Participants received a bolus of glucose at Time Zero, then a bolus of insulin 20 minutes later. Blood was collected through an IV catheter at multiple time points over the course of 4 hours. Glucose and Insulin levels will be plotted on a time course curve and analyzed using the MINMOD algorithm.
Time Frame: week 12
Population: all participants measured
Measure: Mean (Standard Error); unit: [mU/L]^-1 x [min]^-1]
Arm/Group | Fish Oil Group | Control Group
Number analyzed (Participants) | 19 | 14
[mU/L]^-1 x [min]^-1] | 1.7 (.3) | 1.5 (0.2)
Statistical Analysis 1: Comparison: Fish Oil Group vs Control Group; Test type: Superiority; p = 0.5, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Fish Oil Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/14
Other Adverse Events (participants affected / at risk) | 0/19 | 0/14

LIMITATIONS AND CAVEATS:
Study not being powered to identify a difference between groups

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes